CLINICAL TRIAL: NCT02271568
Title: Change in Glomerular Filtration Rate and 24 Hours Ambulatory Blood Pressure After Gastric Bypass Surgery Versus Conventional Weight Loss in Morbid Obesity.
Brief Title: Prospective Cohort Study of the Effect of Bariatric/Metabolic Surgery on Morbid Obesity Patients With Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Tae Kyung Ha, Professor, Hanyang University
Other Study IDs: HYUH 2013-07-024-001
Record Dates: First submitted 2014-10-16; First posted 2014-10-22 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obese patients: 15 Obese patients (BMI>30) having one of comorbidity (type 2 diabetes, dyslipidemia, or hypertension) and morbid obese patients (BMI>35) accepted for bariatric surgery.
  Interventions: Procedure: Bariatric surgery
- Control patients: 15 matched controls receiving Intensive medical therapy
  Interventions: Other: Intensive medical therapy

INTERVENTIONS:
Procedure: Bariatric surgery — Laparoscopic or Robot R-Y gastric bypass
  Groups: Obese patients
Other: Intensive medical therapy — intensive medical therapy according to published guidelines by ADA and EASD
  Groups: Control patients

SUMMARY:
The purpose of this study is to determine the change in kidney function and blood pressure after gastric bypass versus conventional medical therapy in morbid obesity. The study mainly focus on glomerular filtration rate(GFR) with known relation to the renal function and 24 hours ambulatory blood pressure monitoring after intervention of gastric bypass or medical treatment.

DETAILED DESCRIPTION:
Metabolic syndrome is strongly associated with obesity and the patients with this syndrome are at increased risk for cardiovascular disease.

Obesity constitutes a strong risk factor for the development of chronic kidney disease. Among diabetics, obesity is known to amplify the risk for kidney disease.

Bariatric surgery has yielded dramatic results including longitudinal loss of excess body weight and either complete reversal or significant improvement of several features of metabolic syndrome. In addition, many observational studies have demonstrated significant reduction in proteinuria after bariatric surgery.

However, the changes in the component of cardiovascular problem among metabolic syndrome and changes in renal filtration function or progression to end stage kidney disease in morbidly obese patients after weight loss surgery have not been extensively studied. Therefore, our study mainly focus on glomerular filtration rate(GFR) with known relation to the renal function and 24 hours ambulatory blood pressure monitoring after intervention of gastric bypass or medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity (BMI>30) patients with one of comorbidity (type 2 diabetes, dyslipidemia, or hypertension)
* Morbid obese patients (BMI>35)

Exclusion Criteria:

* Prior bariatric surgery
* Malignancy (any type)
* End stage renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 15 Obese patients (BMI>30) having one of comorbidity (type 2 diabetes, dyslipidemia, or hypertension) and morbid obese patients (BMI>35) accepted for bariatric surgery. 15 matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Glomerular filtration rate | prior to surgery - 1, 3, 6, 12month after surgery

SECONDARY OUTCOMES:
Change in excessive body weight | 1, 3, 6, 12month after surgery
Echocardiographic parameter (Systolic and Diastolic parameters, baPWV and LV function) | Before and 12month after surgery
24 hours ambulatory blood pressure | prior to surgery - 1, 3, 6, 12month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyung Ha, MD, PhD, Principal Investigator — Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seongdong-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided